CLINICAL TRIAL: NCT00715455
Title: Phase 2a, Multi-Center, Open Label, Randomized, Feasibility/Safety Study Comparing REG1 Anticoagulation System With Unfractionated Heparin in Subjects Undergoing Elective PCI After Pretreatment With Clopidogrel and Aspirin
Brief Title: Feasibility and Safety Study Comparing REG1 Anticoagulation System With Unfractionated Heparin in Elective PCI
Acronym: REVERSAL-PCI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regado Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REG1-CLIN210
Record Dates: First submitted 2008-02-14; First posted 2008-07-15 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Coronary Artery Disease
Keywords: CAD; PCI; ANTICOAGULANT
MeSH Terms: conditions — Coronary Artery Disease | interventions — Heparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Unfractionated Heparin (Active Comparator): Unfractionated Heparin
  Interventions: Drug: Unfractionated Heparin
- REG1 Partial Rev. (Experimental): REG1 with partial reversal
  Interventions: Drug: REG1
- REG1 Total Rev. (Experimental): REG1 with total reversal
  Interventions: Drug: REG1

INTERVENTIONS:
Drug: REG1 — ii. The REG1 anticoagulation system consists of a drug (RB006) and antidote (RB007). The drug (RB006) is administered via IV bolus to achieve anticoagulation. The antidote (RB007) is administered as an IV bolus dose at approximately 10% the total reversal dose followed by the remaining dose several hours later to counteract RB006 induced anticoagulation.
  Arms: REG1 Partial Rev.
Drug: REG1 — ii. The REG1 anticoagulation system consists of a drug (RB006) and antidote (RB007). The drug (RB006) is administered via IV bolus to achieve anticoagulation. The antidote (RB007) is administered as an IV bolus dose at 100% of the total reversal dose to counteract RB006 induced anticoagulation.
  Arms: REG1 Total Rev.
Drug: Unfractionated Heparin — Heparin will be administered per standard of care at sites
  Other Names: UFH
  Arms: Unfractionated Heparin

SUMMARY:
The purpose of this study is to determine if it is feasible and safe to use the REG1 Anticoagulation System instead of unfractionated heparin during percutaneous coronary intervention (PCI) in subjects with coronary artery disease (CAD).

DETAILED DESCRIPTION:
The study drug, REG1, is the first specific, direct-acting, antidote-controlled anticoagulant ever described. Regado is developing REG1 for use in patients suffering from acute coronary syndrome who undergo coronary revascularization procedures. These procedures, which include coronary artery bypass grafting (CABG) and percutaneous coronary intervention (PCI), put patients at high risk for therapy-related bleeding complications. REG1 is being developed initially to increase therapeutic flexibility and improve patient outcomes in coronary revascularization procedures.

REG1 is a two-component system, consisting of an aptamer-based anticoagulant and its matched antidote. The REG1 anticoagulant component (RB006) is a single-stranded, nucleic acid aptamer. RB006 selectively and potently binds to and inhibits Factor IXa, a protein critical to blood coagulation. The antidote component, RB007, is a complementary nucleic acid that binds to and neutralizes RB006. The binding of RB007 to RB006 causes the predictable and rapid reversal of the RB006 effect and allows the patient's blood to return to normal.

ELIGIBILITY:
Inclusion Criteria:

* Males or females scheduled for non-urgent elective PCI (who do not have certain cardiac parameters) and have not been treated with UHF prior to PCI.
* Subject able to give informed consent and comply with the protocol.
* Negative urine pregnancy test or documented surgical sterilization or menopausal.

Exclusion Criteria:

* Subject weight >120 kg.
* Recent acute coronary syndrome with elevated cardiac markers or ST segment depression at rest.
* Evidence of clinical instability
* Angiographic high-risk.
* A contraindication to anticoagulation or increased risk of bleeding.
* Use of prohibited medications or investigational drugs prior to the study.
* Clinically significant abnormal laboratory findings.
* Planned use of femoral sheath greater than a certain size.
* Known allergy or intolerance to drugs mandated by the study.
* Use of devices other than angioplasty balloons and coronary stents.
* A history of licit drug abuse or illicit drug use or current evidence of such abuse.
* Any other factor that the Investigator feels would put the subject at increased risk if participating in the protocol.
* Lactation.
* Currently enrolled in this or another clinical trial (with some exceptions).
* Participation in an investigational drug or device trial in the past 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Major bleeding using the ACUITY bleeding criteria | until hospital discharge or 48 hours whichever occurs first
Composite of death, nonfatal myocardial infarct (MI), and urgent target vessel revascularization (TVR) | through Day 14 (+/- 3 days)

SECONDARY OUTCOMES:
Angiographic complications | through Day 14 (+/- 3 days)
Femoral Sheath Complications | until the sheath is pulled

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - The Care Group, LLC, Indianapolis, Indiana
  - Henry Ford, Detroit, Michigan
  - UNC, Chapel Hill, North Carolina
  - Geisinger, Danville, Pennsylvania
  - Black Hills Clinical Research Center, Rapid City, South Dakota
- H. Italiano, Buenos Aires, Argentina

REFERENCES:
- [Result] Cohen MG, Purdy DA, Rossi JS, Grinfeld LR, Myles SK, Aberle LH, Greenbaum AB, Fry E, Chan MY, Tonkens RM, Zelenkofske S, Alexander JH, Harrington RA, Rusconi CP, Becker RC. First clinical application of an actively reversible direct factor IXa inhibitor as an anticoagulation strategy in patients undergoing percutaneous coronary intervention. Circulation. 2010 Aug 10;122(6):614-22. doi: 10.1161/CIRCULATIONAHA.109.927756. Epub 2010 Jul 26. PMID 20660806
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581